CLINICAL TRIAL: NCT00256503
Title: Sleep Homeostasis in Primary Insomnia Following Behavioral Treatment
Brief Title: Sleep Homeostasis in Primary Insomnia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: American Academy of Sleep Medicine (Other)
Responsible Party: Principal Investigator, Wilfred Pigeon, PhD, Associate Professor, University of Rochester
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 33-CA-05; 012331 (Other Grant/Funding Number: American Sleep Medicine Foundation)
Record Dates: First submitted 2005-11-16; First posted 2005-11-21 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2016-01

CONDITIONS: Primary Insomnia
Keywords: Primary Insomnia; Insomnia; Sleep
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Insomnia (Experimental): Insomnia subjects who receive 8 session cognitive behavioral therapy for insomnia.
  Interventions: Behavioral: Cognitive-Behavioral Therapy for Insomnia
- Good Sleeper (No Intervention): Good sleeper controls who receive no intervention

INTERVENTIONS:
Behavioral: Cognitive-Behavioral Therapy for Insomnia — Insomnia Subjects receive CBT-I
  Other Names: Insomnia Subjects receive CBT-I
  Arms: Insomnia

SUMMARY:
About 10% of the population is believed to suffer from Primary Insomnia. It is also believed that people with chronic insomnia have a sleep system that is essentially out of alignment (we call this "homeostatic dysregulation"). We also know that a certain form of non-medication therapy called cognitive-behavioral therapy is a very effective treatment for insomnia. It is not known, however, whether cognitive-behavioral therapy actually works by bringing the brain's sleep system back into alignment ("sleep homeostasis"). One of the methods used to measure sleep homeostasis is to observe a person's brain waves during sleep and particularly during sleep that follows a period of sleep loss.

The purposes of this study are to first learn whether persons with insomnia do have a misaligned sleep system compared to persons who do not have insomnia by assessing the sleep of people before and after a period of extended sleep loss. Second, the study will determine whether cognitive-behavioral therapy can re-regulate the sleep system and its response to sleep loss. Third, the final purpose is to examine whether the immune system of people with insomnia is more altered following sleep loss than in the comparison group and whether cognitive-behavioral therapy can alter immune function.

DETAILED DESCRIPTION:
Despite the magnitude of the problem of Primary Insomnia, and the good efficacy of Cognitive Behavioral Treatment for Insomnia (CBT-I), little is known about the pathophysiology of insomnia or whether treatment alters the factors that are thought to maintain chronic insomnia. Three main factors have been explored as contributing to chronic insomnia: hyperarousal, circadian dysrhythmia, and homeostatic dysregulation. Most of the empirical work has been related to the role of hyperarousal along three dimensions: somatic, cognitive, and cortical.

The present study is focused on homeostatic abnormalities and secondarily on hyperarousal as exhibited in subjects with Primary Insomnia (PIs) compared to Good Sleeper controls (GSs). Homeostatic abnormalities will be assessed by evaluating how patients with insomnia respond to sleep deprivation.

This study will use a Modified Sleep Deprivation and Multiple Sleep Latency Test (MSD/MSLT) procedure. Response to the procedure will be assessed in terms of sleep continuity, sleep architecture and electroencephalographic (EEG) power spectral changes during recovery sleep. Hyperarousal will be evaluated using serial measures of somatic (cortisol) and cortical (EEG Beta/Gamma activity) arousal across the sleep deprivation protocol.

These parameters will be evaluated both prior to and following CBT-I in PIs and following an equivalent time interval in GSs.

ELIGIBILITY:
Inclusion Criteria:

Primary Insomnia (PI) subjects:

* Difficulty falling or staying asleep for 6 or more months as evidenced by (a) 30 or more minutes to fall asleep on 3 or more nights per week, or (b) early morning awakenings > 30 minutes prior to desired rise time on 3 or more nights per week
* Reported impaired daytime function attributed to insomnia

Good-Sleeper (GS) controls:

* No history of sleep disorders
* No current sleep complaints and/or complaints of daytime fatigue or sleepiness
* Sleep characterized as restorative and relatively "unperturbable"; and will be defined as: 5-15 minutes to fall asleep and no more than two awakenings per night of > 5 minutes duration

Exclusion Criteria:

* Significant medical or psychiatric illness
* Diagnosed or occult sleep disorders (evident on screening PSG) other than PI
* Hearing or memory impairments
* Non-fluency in spoken or written English
* History of head injury (w/ loss of consciousness) or seizures
* Prescription medication or recreational drug use within 4 weeks of laboratory study
* Tobacco use or consume more than 3 cups of coffee per day (or an equivalent dose of caffeine)

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2005-12; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Slow Wave Sleep (SWS) | Baseline to end of Study (up to 12 weeks)
  Mean minutes of slow wave sleep as measured by standard sleep stage scoring

SECONDARY OUTCOMES:
Delta Power | Baseline to end of study (up to 12 weeks)
  Mean relative power of delta frequency activity during sleep as measured by power spectral analysis

CONTACTS AND LOCATIONS:
Overall Officials: Wilfred R. Pigeon, Ph.D., Principal Investigator — University of Rochester; Michael L. Perlis, Ph.D., Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States